CLINICAL TRIAL: NCT07245979
Title: Assessment of the Effect of Sirtuin Activator Supplementation on Cellular, Metabolic and Anthropometric Parameters in Women
Brief Title: Supplementation With Sirtuin Activators in Women With Increased Body Weight
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Life Sciences (Other)
Collaborators: Poznan University of Medical Sciences (Other); Nutropharma sp. z o.o. (Unknown)
Responsible Party: Principal Investigator, Agata Chmurzyńska, Professor, Poznan University of Life Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Sirt activators
Record Dates: First submitted 2025-10-02; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Obesity & Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: sirtuin activators (Experimental): Sirtuin activators supplementation for 6 months, daily dose of 1278 mg, taken twice a day in a capsulated form. One capsule will contain: resveratrol - 500 g, leucin - 467 mg, Epigallocatechin gallate - 100 mg, quercetin - 100 mg, curcuminoids - 100 mg, niacin 10.7 g. Daily number of capsules will be 2 x 2 = 4.
  Interventions: Dietary Supplement: Sirtuin activators
- Placebo comparator: placebo (Placebo Comparator): Placebo will be an inactive substance (maltodextrin) provided in the same-looking capsules as sirtuin activators. Placebo will be administered twice a day, daily number of capsules will be 2 x 2 = 4.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Sirtuin activators — Sirtuin acitivators supplementation for 6 months
  Arms: Experimental: sirtuin activators
Dietary Supplement: Placebo — Placebo supplementation for 6 months
  Arms: Placebo comparator: placebo

SUMMARY:
The goal of this clinical trial is to learn if the six-month supplementation with sirtuin activators can affect metabolism in 40-to-65-year old women with increased body weight. The main questions it aims to answer are:

Does sirtuin activators affect lipid and carbohydrate metabolism? Does sirtuin activators affect oxydative stress, immune functions and cell ageing?

Researchers will compare sirtuin activators to a placebo (a look-alike substance that contains no drug) to see if drug sirtuin activators works to improve metabolic status.

Participants will:

Take sirtuin activators or a placebo every day for 6 months. Visit the university once every 3 months for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

* females
* age: 40-65 years
* overweight or obese: BMI >25 kg/m2

Exclusion Criteria:

* males
* BMI < 25 kg/m2
* sirtuin activators administration for 3 months prior to study
* pregnancy or breastfeeding
* recent dieting or being on calorie restricted diet
* receiving pharmacotherapy to treat obesity, diabetes or hyperlipidemia
* post-bariatric surgery
* diabetes
* cancer
* chronic kidney, liver or autoimmune diseases
* alcohol addiction

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Concentrations of blood lipids | 6 months, two measurements: at month 0 and 6
  Total cholesterol, Triacyglycerols, low density lipoprotein (LDL) cholesterol, high density lipoprotein (HDL) cholesteroll
Blood glucose concentrations | 6 months, two measurements: at month 0 and 6
  Blood glucose concentration
Ageing biomarkers: transcription level of the p16INK4a gene in peripheral blood mononuclear cells | 6 months, two measurements: at month 0 and 6
  transcription level of the p16INK4a gene in peripheral blood mononuclear cells
Ageing biomarkers: telomere lenght | 6 months, two measurements: at month 0 and 6
  telomere lenght measured in DNA isolated from whole blood
Ageing biomarkers: SA beta galactosidase activity | 6 months, two measurements: at month 0 and 6
  SA beta galactosidase activity
Oxidative stress | 6 months, two measurements: at month 0 and 6
  activities of oxidative stress enzymes in blood

SECONDARY OUTCOMES:
Body mass | 6 months, two measurements: at month 0, 3 and 6
  Measured in kg
Body composition | 6 months, two measurements: at month 0, 3 and 6
  Body composition will include percent body fat and lean body mass measured with air displacement plethysmography
Waist and hips circumference | 6 months, two measurements: at month 0, 3 and 6
  Measured in cm
Genotype analyisis of the Sirt1 gene | baseline
  Nucleotite variants at certain genomic position will be analysed

CONTACTS AND LOCATIONS:
Overall Officials: Agata Chmurzynska, Professor, Principal Investigator — Poznan Univeristy of Life Sciences
Locations (1):
- Poznan University of Life Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No